CLINICAL TRIAL: NCT01316120
Title: Randomized Comparison of Vaginal Self Sampling for Human Papillomavirus (HPV) Testing by Standard Versus Dry Vaginal Swabs
Acronym: HPVDry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Isabelle Eperon, medical doctor, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HPVDry
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Human Papillomavirus Infection
Keywords: Self-collected vaginal samples; HPV; HPV self-obtained sample; HPV specimen transport medium
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPV Dry first (Experimental): Randomization will determine the sequence of the two tests, avoiding potential bias that may advantage the "first" test. All specimens will be tested for the same pathogens (HR-HPV) using the same diagnostic tests
  Interventions: Other: Compare different self-obtained specimen for HPV identification
- HPV standard transport medium (Experimental): Randomization will determine the sequence of the two tests, avoiding potential bias that may advantage the "first" test. All specimens will be tested for the same pathogens (HR-HPV) using the same diagnostic tests
  Interventions: Other: Compare different self-obtained specimen for HPV identification

INTERVENTIONS:
Other: Compare different self-obtained specimen for HPV identification — Instructions will be given to the patients by a research nurse and ICF will be obtained. For specimen collection, participants will be instructed to wash their hands before the procedure. Each participant will receive a package containing a specimen collection kit. Recommendations will be to hold the swab by the end of the handle, to insert the swab into the vagina avoiding contact with the external genitalia, rotate 1 round and to replace the swab in a plastic sleeve (v-DRY) or in a tube containing specimen transport medium (v-STM),.
  Arms: HPV Dry first
Other: Compare different self-obtained specimen for HPV identification — Instructions will be given to the patients by a research nurse and ICF will be obtained. For specimen collection, participants will be instructed to wash their hands before the procedure. Each participant will receive a package containing a specimen collection kit. Recommendations will be to hold the swab by the end of the handle, to insert the swab into the vagina avoiding contact with the external genitalia, rotate 1 round and to replace the swab in a plastic sleeve (v-DRY) or in a tube containing specimen transport medium (v-STM),.
  Arms: HPV standard transport medium

SUMMARY:
Human papillomavirus (HPV) assays are likely to be used in cervical cancer screening. Our objective is to simplify the method of collection of female genital tract specimens by determining if vaginal dry swabs are as accurate as the standard transport medium for HPV diagnosis.

DETAILED DESCRIPTION:
High-risk human papillomavirus (HR-HPV) infections in women are clinically important because they have been associated with nearly all cases of preinvasive and invasive cervical neoplasia1. Genital HR-HPV related infection is common, affecting approximately 10-25% of women, depending on the population and age-groups studied2-4.

With the advance in our understanding of HPV biology and the development of technologies for HPV detection together with the poor sensitivity of a single Pap test, there has been now a growing interest concerning the potential use of HPV DNA testing as a screening tool for cervical cancer5.

Currently, there is no consensus on which sampling method is the most effective for HPV DNA testing. These last years, studies have reported that samples provided by women themselves were suitable for DNA testing and support the feasibility of self-collection for HPV DNA testing6-8. Data from these studies support that it is acceptable for the women and demonstrated that a fairly high concordance rate between the self- and physicians testing method has been achieved.

Potential advantage of self-collection is that it could improve access to health care, reduce healthcare costs and save time for patients and providers. Available data have been reported with the use of specimen transport medium (STM), but the use of dry vaginal swab may potentially offer similar reliability than standard STM. Small studies suggest that HPV test (PCR) sampled by physicians using dry vaginal swab seems to be as accurate as those performed in a standard medium for HPV detection9,10. Dry vaginal swab offers potential advantages in terms of being more convenient for collection and is less expensive than a vaginal swab placed in a transport medium.

The aim of our study is to assess the performance of self-obtained v-DRY versus "standard" v-STM and its acceptability.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older,
* First consultation in our colposcopy unit,
* Understands study procedures and accepts voluntarily to participate by signing the informed consent form (ICF).

Exclusion Criteria:

* Previous hysterectomy,
* Pregnant,
* Virgin,
* Not able to comply with the protocol study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To assess sensibility and specificity of dry swabs for HPV diagnosis | day 1
  Agreement between collection methods in terms of HPV risk categories will be measured using the kappa statistic ( ) with a precision of 10% (95% confidence interval). This measure of agreement is 0 when the amount of agreement is what would be expected by chance and 1 when there is perfect agreement.

SECONDARY OUTCOMES:
Preference about HPV self-collection | day 1
  Women will complete a self administered questionnaire on demographics and preference for sampling method (Dry versus standard)
Sensitivity and specificity of specimen transport medium (STM) | day 1
  Sensitivity and specificity to detect high-risk HPV using v-STM as gold standard will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Petignat, Prof, Study Director — HUG

REFERENCES:
- [Derived] Eperon I, Vassilakos P, Navarria I, Menoud PA, Gauthier A, Pache JC, Boulvain M, Untiet S, Petignat P. Randomized comparison of vaginal self-sampling by standard vs. dry swabs for human papillomavirus testing. BMC Cancer. 2013 Jul 22;13:353. doi: 10.1186/1471-2407-13-353. PMID 23875668